CLINICAL TRIAL: NCT03599921
Title: Treatment Outcome in Eating Disorders
Status: Completed | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Sarah Eckhardt, Principal Investigator, Children's Hospitals and Clinics of Minnesota
Other Study IDs: 47919
Record Dates: First submitted 2018-05-18; First posted 2018-07-26 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Eating Disorder
Keywords: Family-based Treatment; Enhanced Cognitive Behavioral Therapy; Anorexia Nervosa; Other Specified Feeding or Eating Disorder; Bulimia Nervosa; Unspecified Feeding or Eating Disorder; Avoidant/Restrictive Food Intake Disorder; Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Labs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Family-based Treatment: Participants will receive family-based treatment.
  Interventions: Behavioral: Family-based treatment
- Enhanced Cognitive behavioral therapy: Participants will receive enhance cognitive behavioral therapy.
  Interventions: Behavioral: Enhanced Cognitive behavioral therapy
- Family-based Treatment for ARFID: Participants will receive family-based treatment modified for Avoidant/Restrictive Food Intake Disorder (ARFID).
  Interventions: Behavioral: Family-based treatment modified for ARFID
- FBT + UP for ARFID: Participants will receive family-based treatment with the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents, named FBT + UP for ARFID.
  Interventions: Behavioral: FBT + UP for ARFID

INTERVENTIONS:
Behavioral: Family-based treatment — Family-based treatment, or FBT, is the leading evidenced based therapy for children and adolescents with an eating disorder.
  The treatment is a talking type of treatment that involves the whole family and primarily focuses on helping parents play an active and positive role in helping to restore the patient's weight, then hand control of eating back to the patient as is age appropriate. Toward the end of treatment, it is concerned with developmental issues that may have been impacted by the illness.
  Groups: Family-based Treatment
Behavioral: Enhanced Cognitive behavioral therapy — Enhanced Cognitive behavioral therapy, or CBT-E, is a leading evidence based treatment for adolescents and adults with an eating disorder.
  The treatment is a one-to-one talking type of treatment that primarily focuses on what is keeping the eating problem going. It is therefore mainly concerned with the present and the future. It addresses the origins of the problem as needed.
  Groups: Enhanced Cognitive behavioral therapy
Behavioral: Family-based treatment modified for ARFID — Family-based treatment modified for individuals with an ARFID diagnosis is a proposed therapy for treating ARFID.
  The treatment is a talking type of treatment that involves the whole family and primarily focuses on helping parents play an active and positive role in helping to restore patient's weight and variety in eating, as needed.
  Groups: Family-based Treatment for ARFID
Behavioral: FBT + UP for ARFID — Family-based treatment combined with the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents is a proposed therapy for treating ARFID.
  The treatment is a talking type of treatment that involves the whole family and begins with focus on psychoeducation, family engagement, and weight gain as needed. The Unified Protocol is then added to build skills that empower the patient to cope with difficult emotions, address avoidance, and increase tolerance of emotions or disgust responses.
  Groups: FBT + UP for ARFID

SUMMARY:
Do the current eating disorder treatments, i.e., Family-based Treatment (FBT) and Enhanced Cognitive behavioral therapy (CBT-E), offered at the Center for the Treatment of Eating Disorders (CTED) demonstrate effectiveness? Specifically, which type of treatment is most effective for which diagnoses? Participants with Anorexia Nervosa (AN), Bulimia Nervosa (BN), Other Specified Feeding or Eating Disorder (OSFED), or Unspecified Feeding or Eating Disorder (UFED) in this study will self select one of the two treatment groups, FBT or CBT-E.

Additionally, does Family-based Treatment (FBT) modified for Avoidant/Restrictive Food Intake Disorder (ARFID) and Family-based Treatment (FBT) combined with the Unified Protocol (UP) for Transdiagnostic Treatment of Emotional Disorders (FBT+UP for ARFID) demonstrate effectiveness for patients with an Avoidant/Restrictive Food Intake Disorder (ARFID) diagnosis?

DETAILED DESCRIPTION:
Given a significant number of patients who presented for treatment at the Center for the Treatment of Eating Disorders (CTED) and were enrolled in this effectiveness study met criteria for a diagnosis of Avoidant/Restrictive Food Intake Disorder (ARFID), and because there are currently no randomized control trials systematically evaluating children/adolescents with ARFID, a secondary aim was added to this study.

The secondary aim will evaluate the preliminary effectiveness of two treatment groups including: Family-based Treatment (FBT) modified for ARFID and Family-based Treatment (FBT) combined with the Unified Protocol (UP) for Transdiagnostic Treatment of Emotional Disorders (FBT+UP for ARFID) for ARFID patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 6 years of age, attending the CTED clinic for outpatient treatment of a Diagnostic and Statistical Manual, 5th Edition (DSM-5) diagnosed eating disorder in order to be included in this study.

Exclusion Criteria:

* Participants who are receiving inpatient services only and will not return to CTED for outpatient treatment.
* Participants with a co-morbid medical disorder known to influence eating or weight.
* Participants presenting with a significant psychotic disorder.
* Participants who are acutely suicidal.
* Participants who demonstrate significant substance abuse and/or substance dependence.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators plan to enroll 1000 patients, both male and female, ages 6 to adult (18 and older) over a 5 year period. Patients who have been given a Diagnostic and Statistical Manual, 5th Edition (DSM-5) eating disorder diagnosis, and who are seeking outpatient treatment will all be approached for consent to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Therapy effectiveness | Measured at end of treatment (an average of 6-9 months) and at 6 and 12 month follow-up.
  1) Evaluate which therapies work effectively for the treatment of eating disorders, and which types of treatments are most effective for specific diagnoses.

SECONDARY OUTCOMES:
Treatment moderators | Measured at end of treatment (an average of 6-9 months) and at 6 and 12 month follow-up.
  1) Explore predictors and moderators of treatment outcome.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Grange D, Eckhardt S, Dalle Grave R, Crosby RD, Peterson CB, Keery H, Lesser J, Martell C. Enhanced cognitive-behavior therapy and family-based treatment for adolescents with an eating disorder: a non-randomized effectiveness trial. Psychol Med. 2020 Dec 3;52(13):1-11. doi: 10.1017/S0033291720004407. Online ahead of print. PMID 33267919